CLINICAL TRIAL: NCT03006380
Title: Prophylactic Oxytocin Before Versus After Placental Delivery to Reduce Blood Loss in Vaginal Delivery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, AMR HELMY YEHIA, Associate Professor of obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: oxytocin
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxytocin before placental delivery (Experimental): patients who will receive 10 IU of oxytocin (syntocinon®, NOVARTIS, Egypt) intramuscularly at delivery of anterior shoulder of the fetus and an identical placebo injection (normal saline, NACL 0.9%) intramuscularly following delivery of the placenta.
  Interventions: Drug: oxytocin
- oxytocin after placental delivery (Experimental): patients who will receive placebo injection (normal saline, NACL 0.9%) intramuscularly at delivery of anterior shoulder of the fetus and 10 IU of oxytocin (syntocinon®, NOVARTIS, Egypt) intramuscularly following delivery of the placenta.(opposite medication sequence)
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin — Ecbolic used to reduce blood loss
  Other Names: Syntocinon®, NOVARTIS, Egypt

SUMMARY:
Randomized controlled study to assess the efficacy and safety of the timing of administration of prophylactic oxytocin via intramuscular route (before compared to after placental delivery) on blood loss in vaginal delivery.

DETAILED DESCRIPTION:
400 patients will be recruited for the study,Informed consent will be obtained from all patients following the research criteria once they are admitted in active labor, but they will be enrolled and randomized only when they reach the second stage of labor (fully dilated cervix) as it will be difficult in this stage to counsel patients.

The recruited patients will be subjected to the following:

* History taking: with particular emphasis on past medical history (especially for bleeding tendency), past obstetric history.
* Checking vital signs, General and abdominal examination.
* laboratory investigations: complete blood count (CBC)
* Findings of the initial obstetric evaluation follow up, labor duration and the need for oxytocin augmentation will be recorded through a partogram.
* All deliveries will be attended by a senior resident in the hospital.
* Included patients will receive the medication according to randomization tables.
* After allocation, patients will be excluded only if they required cesarean section, instrumental delivery or had multiple or deep vaginal tears that compromise estimation of uterine blood loss.
* All patients will undergo gentle traction to the umbilical cord while providing counter traction against the uterine fundus after signs of placental separation; appearance of bleeding, elongation of the cord.
* All patients will undergo cord clamping and cutting within 30 seconds of delivery.
* All patients will undergo uterine massage for 30 seconds after placental delivery.
* Vital signs (blood pressure and pulse) will be checked 15 minutes, 1 hour and 6 hours after placental delivery.
* CBC will be collected 6 hours after delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Multiparous women (had previous one, up to four deliveries)
2. Term pregnancy (37 completed weeks at least).
3. Singleton viable cephalic pregnancy.
4. Vaginal delivery.

Exclusion Criteria:

1. Primigravida.(first pregnancy)
2. Grand multiparous. (had previous 5 or more deliveries)
3. Maternal illness (involving pregnancy induced condition; PIH,GDM or chronic medical condition; hypertension, cardiac , renal problems)
4. Previous cesarean section, uterine surgery.
5. Patients with bleeding tendency.
6. Previous history of Ante-partum hemorrhage.
7. Previous history of postpartum hemorrhage.
8. Abnormal site of the placenta (detected by ultrasound)
9. Macrosomic baby (EFW more than 4000 gm estimated clinically or by ultrasound)
10. polyhydramnios.(detected by ultrasound)
11. Multiple gestation.
12. Chorioamnionitis.
13. Suspected fetal problem(anomaly, distress)
14. Instrumental delivery.
15. Multiple or deep vaginal tears that compromise the estimation of uterine blood loss.
16. Cesarean delivery

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
blood loss in vaginal delivery | blood loss in the third stage of labor (Up to 60 min after delivery of the baby)

SECONDARY OUTCOMES:
primary postpartum hemorrhage | within 24 hours after delivery
changes in hemoglobin and hematocrit | before delivery and after 6 hours
retained placenta | more than 30 minutes after delivery
length of 3rd stage of labor | Up to 60 min from delivery of baby till delivery of placenta
manual removal of the placenta | if not separated after 30 minutes from delivery
blood pressure | to be measured before delivery after 15 minutes,1 hour,6 hours
maternal pain | during third stage of labor
maternal nausea and vomiting | during 3rd stage of labor
secondary postpartum hemorrhage | after 24 hours and before 6 weeks from delivery
surgical intervention to stop the bleeding | within 24 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Amr Yehia, MD, MRCOG, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided